CLINICAL TRIAL: NCT07228559
Title: A Phase 1b Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of a Suprachoroidal Injection of Avoralstat In Participants With Diabetic Macular Edema
Brief Title: A Study of Avoralstat In Participants With Diabetic Macular Edema
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX4161-111
Record Dates: First submitted 2025-09-26; First posted 2025-11-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Macular Edema (DME)
Keywords: single ascending dose; safety; pharmacokinetics; suprachoroidal injection
MeSH Terms: interventions — avoralstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single dose suprachoroidal injection of avoralstat (Experimental)
  Interventions: Drug: avoralstat

INTERVENTIONS:
Drug: avoralstat — BCX4161 for suprachoroidal injection

SUMMARY:
The goal of this study is to assess the safety and therapeutic potential of a single dose of avoralstat in adult participants with DME.

DETAILED DESCRIPTION:
Study BCX4161-111 is an open-label, single ascending dose study with 24 weeks follow-up in participants with DME. Three cohorts with a minimum of 3 participants enrolled in each cohort with 3 dose levels of avoralstat (low, medium, high) are planned.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female aged 18 years or older
2. Glycated hemoglobin A (HbA1c) < 10% at screening
3. Diagnosis of DME with center involvement requiring medical treatment within 6 months of screening and decreased visual acuity attributable to DME
4. Mild-to-severe non-proliferative diabetic retinopathy (NPDR) with DRSS < 61 in the study eye at screening
5. BCVA between 35 and 80 ETDRS letters (20/25 to 20/200 Snellen equivalent), inclusive, in the study eye at screening
6. CST measured by Heidelberg OCT between 325 and 600 μm in the study eye at screening

Key Exclusion Criteria:

1. Participants who have previously received more than 3 anti-VEGF injections
2. Any history of retinal surgery or other surgical intervention for diabetic ocular complications or anticipated need for use of laser photocoagulation course of any of the procedures listed in the criteria in the study eye during the study period
3. Current medically untreated diabetes mellitus or previous medically untreated diabetes mellitus with initiation of oral or injectable anti-diabetic medication ≤ 3 months prior to screening
4. Active intraocular or periocular infection or active intraocular inflammation in the study eye
5. Intraocular surgery ≤ 3 months prior to screening or anticipated need for ocular surgery in the study eye during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of avoralstat in participants with DME. Incidence and severity of ocular (study eye) and systemic treatment emergent adverse events (TEAEs). | From screening through EOS (Week 24)

SECONDARY OUTCOMES:
Therapeutic potential of avoralstat in participants with DME. Trends in central subfield thickness (CST) as assessed by spectral domain optical coherence tomography (SD-OCT). | From baseline through Weeks 12 and 24
Therapeutic potential of avoralstat in participants with DME. Trends in Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA). | From baseline through Weeks 12 and 24

CONTACTS AND LOCATIONS:
Locations (8):
- United States (3):
  - Investigative Site 6, Sacramento, California
  - Investigative Site 7, Katy, Texas
  - Investigative Site 8, The Woodlands, Texas
- Australia (5):
  - Investigative Site 1, Sydney, New South Wales
  - Investigative Site 2, Sydney, New South Wales
  - Investigative Site 3, Sydney, New South Wales
  - Investigative Site 4, Adelaide, South Australia
  - Investigative Site 5, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No